CLINICAL TRIAL: NCT04207411
Title: Efficacy of Repeated Locoregional Anesthetics Blocks With Bupivacaine in Patients Suffering of Chronic Dentoalveolar Pain. (BADDAP)
Brief Title: Efficacy of Repeated Locoregional Anesthetics Blocks With Bupivacaine in Patients Suffering of Chronic Dentoalveolar Pain.
Acronym: BADDAP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RBHP 2018 MELIN (BADDAP); 2018-002825-49 (EudraCT Number)
Record Dates: First submitted 2019-12-06; First posted 2019-12-20 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2019-12

CONDITIONS: Pain
Keywords: Persistent dentoalveolar pain; bupivacaine; lidocaine; clinical trial; randomization
MeSH Terms: conditions — Pain | interventions — Bupivacaine; Lidocaine

STUDY DESIGN:
Intervention Model Description: bupivacaine or lidocaine randomized treatment.
Who Masked: Participant, Outcomes Assessor
Masking Description: The dentist will prepare the product in another room, so the patient will not know the type of product used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine (Experimental): The dose received at each injection will be 5 mg. One injection per week will be carried out over 4 consecutive weeks
  Interventions: Drug: Bupivacaine
- Lidocaine (Sham Comparator): The dose received at each injection will be 1.25mg. An injection unique per week will be carried out over 4 consecutive weeks.
  Interventions: Drug: Bupivacaine; Drug: Lidocaine

INTERVENTIONS:
Drug: Bupivacaine — Injection of anesthetics blocks once a week during 4 weeks.
Drug: Lidocaine — Injection of anesthetics blocks once a week during 4 weeks.
  Arms: Lidocaine

SUMMARY:
The aim of this study is to evaluate the efficacy of anesthetic blocks repeated with bupivacaine in the management of patients with persistent dentoalveolar pain. Goals are to improve the understanding of the physiopathological mechanisms of persistent dentoalveolar pain and to highlight predictive criteria for the effectiveness of anesthetic blocks.

DETAILED DESCRIPTION:
This is a proof of concept, randomized, controlled prospective pharmacological trial, single blind, with two parallel arms.

The main objective of the study is to evaluate the efficacy of repeated locoregional anesthetic blocks with bupivacaine in patient's persistent dentoalveolar pain compared to a control group receives a simulated anesthesia (local anesthesia with lidocaine).

The secondary objectives are :

* to evaluate the tolerance of repeated locoregional anesthetic blocks to bupivacaine patients with persistent dentoalveolar pain compared to control receiving simulated anesthesia (local anesthesia with lidocaine).
* to evaluate demographic and nosological predictive factors (age of symptoms, Quantitative Sensory Testing results) and psychometric (anxiety, depression, dramatization) of the effectiveness of anesthetic blocks.

After signing the informed consent, the patients participate will be randomized to anesthetic block treatment with bupivacaine or lidocaine.

During the 1st step of the study patients will participate at 6 visits (day -7, day 0, day 7, day 14, day 21 and M2) and will receive either a series of 4 locoregional anesthetic blocks with bupivacaine or a series of 4 local anesthesia with lidocaine ("simulated" control group) at day 0, day 7, day 14 and day 21. The main criterion is raised 2 months after the end of the series.

During the 2nd step

* The patients from experimental group will be followed until month 6 (2 visits: month 3 month 6).
* The patients from control group :
* will received in open (if they want) a series of 4 locoregional anesthetic blocks with bupivacaine (day56, day,63, day 70, day 77) and will be followed during 6 months after the first injection (7 visits: day 63, day 70, day 77, month 3, month 4, month 5, month 8)
* will be followed until month 6 ((2 visits: month 3 month 6).

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over 18, with persistent dentoalveolar pain defined according to the criteria:

  * daily presence (> 2 hours / day and for more than 3 months) and continues pain;
  * located at one or more teeth or at the level of the alveolar bone;
  * not following a nervous path;
  * clinical, radiological and neurological examinations showing no cause organic visible;
  * dental causes excluded by appropriate tests;
  * local or systemic pathologies related to pain apart.
* Pain intensity greater than or equal to 4/10 on numerical scale
* Patient informed of the constraints of the study and having given his written consent. Benefiting of a social security scheme.
* Mastering correctly French.

Exclusion Criteria:

* Pregnant women, breastfeeding, or likely to be pregnant.
* Oral pain of known origin (cancerous, infectious, traumatic).
* Patient having modified (stopped, started or modified dosage) in the last 2 month local or systemic medication that may interfere with the study results (for example, patients taking long-range psychotropic drugs will not be excluded).
* All medical pathology judged by the investigator as not compatible with the study.
* Known hypersensitivity to local amide-bound anesthetics or to any of the excipients
* Treatment anticoagulant or known disorder of blood
* Porphyria.
* Atrioventricular conduction requiring training permanent electrosystol not yet realized.
* Epilepsy not controlled by a treatment.
* Patient non-cooperating, not speaking or not reading fluently French or in the impossibility of understanding the principle of a pain scale or understanding the study or to sign an informed consent.
* Patient under guardianship, curatorship, or deprived of liberties.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients (with persistent dentoalveolar pain). with at least 30% pain reduction | difference compared to the basal value at day 0 (visit 1) to value at Month 2 (visit 6)
  Mean numerical scale on journal of pain (last 7 days)

SECONDARY OUTCOMES:
Brief Pain Inventory | The questionnaire will be completed at day-7, and month 2 for all patients and then "month 3 and month 6" for patient of experimental group or visit month 4, month 5, month 8 for control group.
  This self-questionnaire will assess the pain intensity and impact of pain on the patient's life. He understands : a body image ; the maximum pain, the weakest pain, the usual pain of the last 15 days (numerical scale 0 to 10); the description of the current analgesic treatment; a assessment of relief by a percentage scale (0 to 100%); the study of the impact of pain on mood, relationships with other people, walking, sleep, work, joy of life, leisure, activities in general (scales numeric, rating from 0 (normal) to 10 (activity impossible).
Patient's Global Impression of Change (PGIC) | The questionnaire will be completed at month 2 for all patients and then "month 3 and month 6" for patient of experimental group or visit month 4, month 5, month 8 for control group.
  Its purpose is to evaluate in a general way the effectiveness of a treatment felt by the patient. This scale consists of 7 levels of descriptors answering the question "Since start of treatment, how would you describe the change (if any) in your limitations of activities, your symptoms, your emotions and your quality of life in general, related to your affection painful? ", Divided according to 3 modalities: improvement: (7) very, (6) medium, (5) slightly, unchanged( 4), worsen (3) slightly, (2) medium, (1) very.
Neuropathic Pain Assessment Questionnaire (QEDN) | The questionnaire will be completed at day-7, and month 2 for all patients and then "month 3 and month 6" for patient of experimental group or visit month 4, month 5, month 8 for control group.
  The Neuropathic Pain Assessment Questionnaire is a self-questionnaire that has been specifically validated to assess and monitor the different aspects of neuropathic pain and is sensitive to change. This questionnaire consists of twelve questions, ten of which relate to the description of pain by measuring its intensity using a numerical scale, that is, by grading the pain from 0 (no pain) to 10 (maximum pain imaginable). The remaining two questions each offer five answers about the duration of spontaneous pain over 24 hours (from "1 to 3 hours per day" to "continuously") and the number of painful seizures (paroxysms) over 24 hours (from "no painful crisis" to "more than 20"). The ten descriptive questions can be grouped into 5 dimensions. The sum of the 10 questions gives the total score scored on 100 and each dimension gives a sub-score.

CONTACTS AND LOCATIONS:
Overall Officials: Céline Melin, BDS, PhD, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No